CLINICAL TRIAL: NCT06522516
Title: A Nurse-led Family-oriented Resilience Program for Caregivers of Community-dwelling Dependent Older Adults: a Three-arm Controlled Trial
Brief Title: A Nurse-led Family-oriented Resilience Program for Caregivers of Community-dwelling Dependent Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Anni Wang, Associate Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: A family resilience program
Record Dates: First submitted 2024-07-20; First posted 2024-07-26 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Caregiver Burden
Keywords: family resilience; caregiver; distress; older adults
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: 2 intervention groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caregiving training group (Experimental): Caregiving training group will receive an evidence-based caregiving training via manual during nurse home visit.
  Interventions: Behavioral: Evidence-based caregiving training; Behavioral: usual service
- Caregiving training plus family resilience group (Experimental): Caregiving training plus family resilience group will receive an evidence-based caregiving training and family resilience psychological intervention via manual during nurse home visit
  Interventions: Behavioral: Evidence-based caregiving training; Behavioral: family resilience intervention; Behavioral: usual service
- Control group (Active Comparator): Controlled group will receive usual community service by nurse.
  Interventions: Behavioral: usual service

INTERVENTIONS:
Behavioral: Evidence-based caregiving training — This is designed based on evidence of daily living activity ability caregiving, including① Dietary training: guiding caregivers to choose appropriate tableware according to the functional status of disabled elderly people, and training them in eating posture such as changing positions and using tableware; ② Dressing training: guide caregivers to train disabled elderly people on how to put on and take off clothes, shoes, socks, etc.; ③ Personal hygiene training: including washing face, hands, brushing teeth, etc.; ④ Excretion function training: including urination function training and defecation function training; ⑤ Mobile training: including support walking training, cane walking training, etc.; ⑥ Wheelchair training: Guide caregivers to use wheelchairs according to the specific situation of disabled elderly people.
  Arms: Caregiving training group; Caregiving training plus family resilience group
Behavioral: family resilience intervention — The intervention will be developed based on the Maccubbin Family Resilience Theory, and Delphi methods. The content will contain 8 topics and be incorporated into caregiving training manual.
  Arms: Caregiving training plus family resilience group
Behavioral: usual service — This means the usual service provided by the local community health center from nurses during bi-weekly home visit.

SUMMARY:
This is a 3-arm controlled trial. The participants are caregivers of the community-dwelling dependent older adults. There will be around 105 participants to be recruited and randomly allocated into 3 groups. Caregiving training group will receive a evidence-based caregiving training delivered via home visit of community nurse. Caregiving training plus family resilience group will additionally receive a structured family resilience intervetion. Control group will receive usual community health care service by nurses. The primary outcomes are caregiving ability, family resilience and psychological distress, and the secondary outcomes are caregiving burden, resilience, coping, social support, and quality of life the caregivers and the older adults. The measurement will be conducted four times at baseline, after, 1-month and 3-month after intervention.

ELIGIBILITY:
Inclusion Criteria:

* ①The degree of disability of the caregiver is moderate to severe activity of daily living score above;

  * The primary caregivers are≥18 years old ;

    * The primary caregivers bear the most important care task during care, and the continuous care time are≥3 months ; -④The psychological pain thermometer score of the primary caregivers are≥5 points (the previous cross-sectional survey results showed that when the psychological pain thermometer score of the primary caregivers in disabled elderly are 5 points, the highest Youden index is obtained, and the sensitivity, specificity, positive predictive value, and negative predictive value are also high. Therefore, participants with scores above 5 points are screened as potential research subjects ); -⑤No cognitive impairment or language expression disorders; -⑥The primary caregivers have smart phones and can use them skillfully, and have access to the Internet; -⑦Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

* ①Currently participating or having received intervention from other healthcare teams within the past three months;

  * There are paid personnel such as nannies participating in the care.

    * Those who voluntarily withdrew from the research process;

      * During the research process, due to significant adverse events (such as death) involving disabled elderly individuals or primary caregivers, they were unable to continue participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
family resilience | There will be 4 measurements, before, immediately after and，1-month, 3-month after the intervention.
  The Walsh Family Resilience Questionnaire Chinese Version (WFRQ-C) is used to measure the level of family resilience of primary caregivers. The questionnaire includes three dimensions and 26 items: family beliefs, communication and resolution, and external support. The questionnaire items are evaluated using a Likert 5-point rating system, with scores ranging from 1 to 5 from "never" to "always". The higher the score, the higher the level of family resilience. The Cronbach's alpha coefficient of the questionnaire is 0.93, with a test-retest reliability of 0.96, indicating good validity.
psychological distress | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  Distress thermometer (DT): used to assess the level of psychological distress of primary caregivers. This scale was designed by Roth and translated into China by Tang Lili et al. in 2011. DT is a visual analog scale scale ranging from 0 to 10 points (0 indicates no psychological distress, 10 indicates extreme psychological distress). The reliability of the Chinese version DT retest is r=0.80, and the calibration validity is good.
caregiving ability | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  Caregiver Task Inventory (FCTI): used to measure the caregiving ability of primary caregivers. This scale consists of 5 dimensions (adapting to caregiver roles, responding to needs and providing assistance, handling personal emotions, evaluating family and community resource professionals, and adjusting life to meet caregiving needs), with a total of 25 items.The total score is 50 points, with higher scores indicating more caregiving difficulties for caregivers. The Cronbach's alpha coefficient of the scale is 0.93, indicating good construct validity.

SECONDARY OUTCOMES:
caregiving burden | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  The Zarit Burden Inventory (ZBI) is used to measure the caregiving burden of primary caregivers. This scale is a self-assessment scale consisting of two dimensions: personal burden and responsibility burden, with a total of 22 items. The Cronbach's alpha coefficient of this scale is 0.87.
resilience | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  The Connor Davidson Resilience Scale (CD-RISC) is used to assess the psychological resilience of primary caregivers.The Chinese version of CD-RISC includes 3 dimensions (resilience, strength, and optimism), 25 items, and is rated on a scale of 1-5, with higher scores indicating higher levels of psychological resilience. The Cronbach's alpha coefficient of the scale is 0.91, indicating good criterion related validity.
coping | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  Simplified Coping Style Questionnaire (SCSQ): used to assess the coping strategies of primary caregivers. This scale was developed by Jie Yaning in 1998. It includes two dimensions (positive coping and negative coping), with 20 items. The positive coping dimension includes items 1-12, and the negative coping dimension includes items 13-20. It is rated on a scale of 0-3 out of 4. The higher the total score of the positive dimension, the more likely the survey respondents are to adopt positive coping methods; The higher the total score of the negative coping dimension, the more inclined the survey respondents are to adopt negative coping strategies. The Cronbach's alpha coefficient of the positive coping style in this scale is 0.89, and the Cronbach's alpha coefficient of the negative coping style is 0.78.
social support | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  Perceived Social Support Scale (PSSS): used to measure the perceived level of social support among primary caregivers. This scale was developed by Zemit in 1987 and later translated into Chinese by Huang Li et al. and introduced into China. This scale consists of 3 dimensions (family support, friend support, and other support), with a total of 12 items. It uses a 7-point scoring system ranging from 1 to 7, with higher total scores indicating higher levels of social support. The Cronbach's alpha coefficient of this scale is 0.92, indicating good test-retest reliability and construct validity.
Quality of life of caregiver | There will be 4 measurements, before, immediately after,1-month, and 3-month after the intervention.
  The European Five Dimensional Five Level (EQ-5D-5L) health scale: used to measure the quality of life of disabled elderly and primary caregivers. This scale was developed by the European Society for Quality of Life and includes a brief descriptive system questionnaire and a visual analog scale. The Cronbach's alpha coefficient of this scale is 0.857, indicating good validity.
Quality of life of older adults | There will be 4 measurements, before, immediately after, 1-month, and 3-month after the intervention.
  The European Five Dimensional Five Level (EQ-5D-5L) health scale: used to measure the quality of life of disabled elderly and primary caregivers. This scale was developed by the European Society for Quality of Life and includes a brief descriptive system questionnaire and a visual analog scale. The Cronbach's alpha coefficient of this scale is 0.857, indicating good validity.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT06522516/Prot_SAP_000.pdf